CLINICAL TRIAL: NCT04419363
Title: 12-months of Treatment With Burosumab in Children and Adolescents With X-linked Hypophosphatemia: a Prospective Longitudinal Cohort Study
Brief Title: Burosumab in Children and Adolescents With X-linked Hypophosphatemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Volha Zhukouskaya, MD, PhD, Bicetre Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200528104746
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Rare Diseases; X-linked Hypophosphatemia
Keywords: X-linked hypophosphataemia; fibroblast growth factor 23; burosumab; hyperparathyroidism
MeSH Terms: conditions — Rare Diseases; Familial Hypophosphatemic Rickets; Hyperparathyroidism | interventions — burosumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The whole cohort (Experimental): Children affected with X-linked hypophosphatemia of average age of 9.8 years were switch from conventional therapy to burosumab
  Interventions: Drug: Burosumab Injection

INTERVENTIONS:
Drug: Burosumab Injection — Children affected with X-linked hypophosphatemia were switched from conventional therapy to burosumab

SUMMARY:
In this prospective longitudinal cohort study we studied the efficacy and safety of burosumab in real-clinical practice for <13- and >13-years old children affected with X-linked hypophosphatemia.

57 children with XLH were switched from conventional treatment to burosumab. After 12 months we assessed the efficacy and safety of treatment with burosumab on the whole cohort and separately on the cohort of >13-years old adolescents.

ELIGIBILITY:
Inclusion Criteria:

* insufficient response or refractory to conventional therapy;
* complications of conventional therapy: hypercalciuria and/or nephrocalcinosis, and/or persistent secondary hyperparathyroidism;
* need for rapid restoration of phosphate metabolism, e.g., late diagnosis (aged >8 years) and/or preparation for planned orthopaedic surgery.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2018-03-18 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2022-09-16 (Estimated)

PRIMARY OUTCOMES:
Radiological changes in rachitic lesions evaluated with knee MRI | 12 months
  maximum width of the physis and transverse extent of widening

SECONDARY OUTCOMES:
serum phosphate | 12 months
  mmol/l
renal phosphate reabsorption | 12 months
  mmol/l
alkaline phosphatase | 12 months
  U/l
1,25(OH)vitaminD | 12 months
  pg/ml
parathyroid hormone | 12 months
  ng/l
height | 12 months
  standard deviation score
functional capacity | 12 months
  6-minute walk test, standard deviation score
incidence of dental abcesses | 12 months
  dental examination
incidence of hearing problems | 12 months
  ORL examination, audiogramm
incidence of neurological problems (craniosynostosis, Chiari I malformation) | 12 months
  neurosurgical examination and brain MRI
incidence of nephrocalcinosis | 12 months
  renal ultrasound
incidence of hyperparathyroidism | 12 months
  blood levels of parathyroid hormone
incidence of any side effects | 12 months
  registration of any side effects during the treatment by telephone call

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Bicetre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No